CLINICAL TRIAL: NCT01051622
Title: An Exploratory SPECT Imaging Study to Assess the Utility of High-specific Activity 99mTc-HMPAO Labeling as a Tool to Detect PBMC and Lymphocyte Trafficking in the Small Bowel or Ileo-caecal Region of Crohn's Disease Patients
Brief Title: PBMC (Peripheral Blood Mononuclear Cells) /Lymphocyte SPECT (Single Photon Emission Computerized Tomography) Imaging in Crohn's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 113265
Record Dates: First submitted 2009-12-03; First posted 2010-01-18 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Crohn's Disease
Keywords: PBMC (Peripheral Blood Mononuclear Cells); Crohn's Disease; SPECT (Single Photon Emission Computerized Tomography)
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PBMC Trafficking (Experimental): In part B, Patients undergo a blood draw (up to150 mL) and the PBMC's are separated and selected or 99mTc-HMPAO labeling. The purified and labelled cells will be re-introduced into the patient by intravenous infusion and one SPECT scan and up to 8 serial planar scintigraphy scans will initially be conducted over up to 6 hours within 1 scan session. All suitable patients showing evidence of cellular uptake in the ileo-caecal region and/or small bowel at Visit 1 will be progressed to an identical second cell labeling and scanning session at Visit 2 (48 hours later). Subjects showing no evidence of cellular uptake in the ileo-caecal region or small bowel at Visit 1 (negative scan) will be withdrawn from the study and proceed to the follow-up.
  Interventions: Other: Labeling Ceretec
- T Lymphocyte Trafficking (Experimental): In part B, Patients undergo a blood draw (up to150 mL) and the T lymphocyte cells are separated and selected or 99mTc-HMPAO labeling. The purified and labelled cells will be re-introduced into the patient by intravenous infusion and one SPECT scan and up to 8 serial planar scintigraphy scans will initially be conducted over up to 6 hours within 1 scan session. All suitable patients showing evidence of cellular uptake in the ileo-caecal region and/or small bowel at Visit 1 will be progressed to an identical second cell labeling and scanning session at Visit 2 (48 hours later). Subjects showing no evidence of cellular uptake in the ileo-caecal region or small bowel at Visit 1 (negative scan) will be withdrawn from the study and proceed to the follow-up.
  visit.
  Interventions: Other: Labeling Ceretec

INTERVENTIONS:
Other: Labeling Ceretec — Technetium-99m is used to radiolabel cells of interest i.e PBMC's

SUMMARY:
Using scintigraphic imaging including planar scintigraphy and SPECT, this study will evaluate the utility of two different ex vivo 99mTc-HMPAO labelled mononuclear cell populations in order to select the optimal methodology (using PBMC or purified lymphocyte subpopulations) for future drug intervention studies in Crohn's disease.

Two parallel exploratory approaches will be investigated to enrich for lymphocyte populations expressing leukocyte trafficking inhibitors. In the first, whole blood will be fractionated on a ficoll gradient to purify a heterogeneous population of all the peripheral blood mononuclear cells (PBMC) for labelling. Secondly, further enrichment will be attempted using depletion of PBMC fractions of monocytes and B cells.

DETAILED DESCRIPTION:
This study is based on the established technology of scintigraphic 'white cell scanning', in which the leukocytes in a limited volume of patient's blood are radiolabeled with indium-111 or technetium-99m, re-introduced into the circulation, and their subsequent trafficking and accumulation in areas of active inflammation is visualised by scintigraphic imaging. This methodology is routinely used for diagnosis of inflammatory conditions and pharmacodynamic changes have been documented in the literature. As it is intended that this technology could be used in future drug intervention studies.

However, because this sub-population labelling methodology remains exploratory, this study will investigate the utility of such techniques for use in future clinical trials in Crohn's patients.

Two parallel exploratory approaches will be investigated to enrich for lymphocyte populations expressing leukocyte trafficking inhibitors. In the first, whole blood will be fractionated on a ficoll gradient to purify a heterogeneous population of all the peripheral blood mononuclear cells (PBMC) for labelling. Secondly, T lymphocytes will be further enriched by depletion of monocytes and B cells from PBMC fractions. In part A one scintigraphy scan will be performed in healthy volunteers to confirm that the purification and labelling procedure does not show abnormal biodistribution compared to the known physiological distribution of labelled mononuclear cells [Bennink, 2008].

In part B, Crohn's disease patients will then be recruited to undergo two scintigraphy scans 48-72 hours apart to establish intra-patient variability and feasibility of the repeated procedure that will be used in subsequent studies for therapeutic intervention. Analysis of SPECT images will be performed using a standardized scoring system.

ELIGIBILITY:
Inclusion

A subject will be eligible for inclusion in this study only if all of the following criteria apply:

Part A only:

1. Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, vital signs, ECG, complete blood count and clinical chemistry. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.

   Part A and B:
2. Male or female over 18 years of age inclusive, at the time of signing the informed consent.
3. A female subject is eligible to participate if she is of:

   • Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<140 pmol/L) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods in Section 8.1 if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.

   Part B only:
4. A history of CD for at least 3 months with a diagnosis confirmed by radiologic, endoscopic or histological assessment.
5. Moderate to severe CD as evidenced by an elevated retrospective CDAI score (of

   ≥150) and 1 or more of the following:
   * CRP (of ≥5 mg/L); or
   * recent (within 4 weeks before the screening visit) evidence of active CD by CT scan, MRI scan or endoscopy. Scans must be part of the patients routine care and should not be conducted as a screening test for this study.
6. Radiographic (barium, CT, MRI) or endoscopic evidence of small bowel involvement (if a patient has had a surgical intervention, evidence of small bowel involvement must have been obtained after the procedure).

Exclusion

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

Part A and B:

1. Known or positive infection with hepatitis B, hepatitis C or HIV.
2. The subject has participated in a clinical trial and has received an investigational product within the following time period prior to Day 1 of the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
3. Previous inclusion in a research and/or medical protocol involving nuclear medicine, PET or radiological investigations with significant radiation burden (a significant radiation burden being defined as ICRP category IIb or above: no more than 10 mSv in addition to natural background radiation, in the previous 3 years including the dose from this study).

   Part B only:
4. Patients with active Crohn's disease with small bowel involvement who are not yet receiving treatment for whom it is judged inappropriate to defer initiating steroid or other treatment for up to 13 days (the maximum interval from screening to last imaging session).
5. Patients who are corticosteroid dependent for whom it is judged inappropriate to defer increasing the dose of steroids or initiating other treatment for up to 13 days (the maximum interval from screening to last imaging session).
6. Patients who are refractory to steroids or immunosuppressants or anti-TNFs for whom it is judged inappropriate to defer change of medical management or surgical intervention for up to 13 days (the maximum interval from screening to last imaging session).
7. The subject is taking >20mg/day Prednisolone or a prednisolone equivalent during the 4 weeks prior to screening
8. The subject received treatment natalizumab within 12 weeks prior to study entry;
9. The subject has Hb<10 g/l or Lymphocyte count <10^9 /l
10. Known C. difficile infection, or a clinical suspicion of a pathogenic bowel infection (including significant infection due to fistula).
11. Suspected or diagnosed intra-abdominal abscess or bowel perforation
12. The subjects has had bowel surgery (other than appendectomy) within 12 weeks prior to randomization or is likely to require abdominal surgery within 1 month of screening
13. Concurrent illness, infection or disability (including malignancies or neoplastic disease of the bowel) that may affect the interpretation of clinical data, or otherwise contraindicates participation in this clinical study (e.g., an unstable cardiovascular, autoimmune, renal, hepatic, pulmonary, endocrine, metabolic, gastrointestinal, hematologic, psychiatric or neurological condition).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-01; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Quantification of scintigraphic activity score for small bowel disease (for both PBMC and lymphocyte imaging methodologies) | 1 day

SECONDARY OUTCOMES:
Tolerability endpoints including AEs | Up to 3 weeks
Variability and reproducibility of the PBMC and lymphocyte imaging methodologies at visits 1 and 2. | Up to 3 days
Rate of label accumulation in small bowel | 1 day
Circulating PBMC and lymphocyte subpopulation cell counts and correlation with scintigraphic activity scores. | 1 day
Correlation between CDAI, CRP, calprotectin, ASCA antibodies and SAS | Up to 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, Leuven, Belgium
- GSK Investigational Site, Amsterdam, Netherlands